CLINICAL TRIAL: NCT05927038
Title: Coffee Consumption, the Gut Microbiome, and the Microbiota-Gut-Brain Axis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Cork (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: APC115
Record Dates: First submitted 2023-05-29; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Healthy
Keywords: Coffee; Microbiome-gut-brain-axis; Prebiotic; Polyphenol; Cognition; Stress; Mood; Behavior; Inflammation; Gut Microbiota; Caffeine
MeSH Terms: conditions — Behavior; Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caffeinated coffee (Experimental): 4 sachets (1.8 grams each) of instant, caffeinated coffee
  Interventions: Other: Caffeinated coffee
- Decaffeinated coffee (Experimental): 4 sachets (1.8 grams each) of instant, decaffeinated coffee
  Interventions: Other: Decaffeinated coffee

INTERVENTIONS:
Other: Caffeinated coffee — After 2 weeks of coffee abstinence (washout), participants who were coffee drinkers were randomly allocated to receive either 4 sachets (1.8g each) of caffeinated instant coffee per day for 3 weeks. Participants were blinded to coffee contents.
  Arms: Caffeinated coffee
Other: Decaffeinated coffee — After 2 weeks of coffee abstinence (washout), participants who were coffee drinkers were randomly allocated to receive either 4 sachets (1.8g each) of decaffeinated instant coffee per day for 3 weeks. Participants were blinded to coffee contents.
  Arms: Decaffeinated coffee

SUMMARY:
The aim of this study is to investigate the potential of coffee to act as a prebiotic to alter gut microbiota and improve mood, memory and cognitive performance.

DETAILED DESCRIPTION:
The aim of this study is to investigate the potential of coffee to act as a prebiotic to alter gut microbiota and improve mood, memory and cognitive performance. Additional gut-brain axis pathways-related parameters such as inflammation, short chain fatty acids and other metabolites production and physiological stress levels will be explored. Moreover, differences between caffeinated and decaffeinated coffee consumption will be investigated to determine whether observed effects are attributed to caffeine or other coffee components.

To determine the mechanism of action underlying the beneficial effects of coffee, coffee drinkers abstained from coffee and caffeine for a 2-week washout period following the baseline visit. Coffee drinkers further underwent an intervention in which they consumed either 4 sachets (1.8 grams each) of instant caffeinated or decaffeinated coffee per day for 3 weeks of using a double-blind, randomised, parallel design. Reaction time, socioemotional processing, visual and episodic memory, learning, and an attentional task were administered to measure cognitive performance. Self-report questionnaires on mood, behavior and lifestyle were administered and response to an acute stressor was assessed. Biological samples of saliva, urine, blood, and stool were collected to investigate microbiome-gut-brain-axis signaling.

ELIGIBILITY:
Inclusion Criteria:

1. Be able to give written informed consent.
2. Be between 30 and 50 years of age.
3. Be in generally good health as determined by the investigator.
4. Drink moderate amounts of coffee daily (3-5 cups/day)

Exclusion Criteria:

1. Are less than 30 and greater than 50 years of age.
2. Have a significant acute or chronic coexisting illness [cardiovascular, gastrointestinal (GI) [to include functional GI disorders, inflammatory bowel disease, coeliac disease, lactose intolerance, food allergies], immunological, psychiatric [to include formal or as determined by MINI Psychiatric interview, diagnosis of current major depression, anxiety disorder, bipolar spectrum disorder, schizophrenia, other DSM-IV Axis I disorder], neurodevelopmental disorders, immunological, metabolic disorders [to include type I or II diabetes], or any condition which contraindicates, in the investigators judgement, entry to the study,
3. Have a condition or taking a medication that the investigator believes would interfere with the objectives of the study, pose a safety risk or confound the interpretation of the study results; all psychoactive medications [to include anxiolytics, antipsychotics, antidepressants, anticonvulsants, centrally acting corticosteroids and opioid pain relievers), laxatives, enemas, antibiotics, anti-coagulants, over-the counter non-steroidal anti-inflammatories (NSAIDS). Subjects should have a wash-out period of 4 weeks.
4. Be hypertensive.
5. Current prebiotic or probiotic supplement use (a wash-out period of 4 weeks after cessation will allow entry to the study), or habitual consumption of foods deemed by the investigator to be particularly rich in prebiotic fibres or probiotic strains or are vegan.
6. Females who are pregnant or planning a pregnancy, or lactating.
7. Participants who are not fluent in English.
8. Participants who have dyslexia or dyscalculia.
9. Are a current habitual daily smoker.
10. Individuals who, in the opinion of the investigator, are considered to be poor attendees or unlikely for any reason to be able to comply with the trial.
11. Subjects receiving treatment involving experimental drugs. If the subject has been in a recent experimental trial, these must have been completed not less than 30 days prior to this study.
12. Have a malignant disease or any concomitant end-stage organ disease.
13. Have already done a study in the lab in the past 4 years

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2021-09-21 (Actual); Primary Completion 2023-01-18 (Actual); Study Completion 2023-01-18 (Actual)

PRIMARY OUTCOMES:
Microbiota composition and function | Differences between groups at baseline, at 2-week coffee abstinence and at 3-week coffee intervention
  Shotgun metagenomics of fecal samples

SECONDARY OUTCOMES:
Gut microbial metabolites (including Short-Chain fatty acids) | Differences between groups at baseline, at 2-week coffee abstinence and at 3-week coffee intervention
  Untargeted metabolomics of fecal samples
Coffee-related metabolites | Differences between groups at baseline, at 2-week coffee abstinence and at 3-week coffee intervention
  Targeted metabolomics of coffee-related metabolomics in fecal and urine samples

OTHER OUTCOMES:
Cognitive performance: attention | Differences between groups at baseline, at 2-week coffee abstinence and at 3-week coffee intervention
  Assessment of attention using the Paced Auditory Serial Addition Test (PASAT)
Cognitive performance - Episodic memory | Differences between groups at baseline and at 3-week coffee intervention
  Assessment of episodic memory using the Modified Rey Auditory Verbal Learning Test (ModRey)
Cognitive performance - Learning and visual memory | Differences between groups at baseline and at 3-week coffee intervention
  Assessment of learning and visual memory using the Paired Associates Learning task
Cognitive performance - Processing speed | Differences between groups at baseline and at 3-week coffee intervention
  Assessment of processing speed using the Motor Screening Test
Cognitive performance - socioemotional processing | Differences between groups at baseline and at 3-week coffee intervention
  Assessment of socioemotional processing using the Emotion Recognition Task
Responses to acute stressor | Differences between groups at baseline and at 3-week coffee intervention
  Self-report mood and cortisol responses to the Socially Evaluated Cold Pressor Test
Inflammatory profile | Differences between groups at baseline, at 2-week coffee abstinence and at 3-week coffee intervention
  Inflammatory markers analysis in LPS-stimulated blood and in the plasma using MSD multiplex technology. The inflammatory markers analyzed were: C-reactive protein, IL6,IL10,IL8, INFgamma, TNFalpha, IL1beta.
Cortisol awakening response | Differences between groups at baseline, at 2-week coffee abstinence and at 3-week coffee intervention
  Cortisol awakening response measurement using ELISAs
Self-reported questionnaires | Differences between groups at baseline, at 2-week coffee abstinence and at 3-week coffee intervention
  Completion of self-reported questionnaires on mood, depression, anxiety, impulsivity, emotional reactivity, stress, and sleep quality. Low scores represents better outcomes.
Genotyping adenosine receptor A2A | At the baseline
  Genotyping of 2 SNPs of the A2A receptor using blood (caffeine is an antagonist of the A2A receptor.

CONTACTS AND LOCATIONS:
Overall Officials: John F Cryan, PhD, Principal Investigator — UCC
Locations (1):
- University College Cork, Cork, Ireland

IPD SHARING:
Plan to Share IPD: No